CLINICAL TRIAL: NCT06192212
Title: Relationship Between Different Nutritional Modalities and Tumor Prognosis After Minimally Invasive Esophagectomy
Brief Title: PPIO-005 The Relationship Between Different Nutritional Pathways and Tumor Outcomes After Minimally Invasive Esophagectomy
Status: Completed | Type: Observational
Sponsor: Daping Hospital and the Research Institute of Surgery of the Third Military Medical University (Other)
Responsible Party: Principal Investigator, WEI GUO, chief physician, Daping Hospital and the Research Institute of Surgery of the Third Military Medical University
Other Study IDs: WeiGuo
Record Dates: First submitted 2023-12-21; First posted 2024-01-05 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Esophageal Squamous Cell Carcinoma
Keywords: esophageal squamous cell carcinomas; Jejunostomy; nutrition; postoperative complications; Anastomotic leak
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma; Postoperative Complications; Anastomotic Leak

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Jejunostomy group: Intraoperative jejunostomy tube placement received
- Non-jejunostomy group: Intraoperative jejunostomy tube placement not received

SUMMARY:
As there is no consensus to date on the optimal postoperative nutritional support route for patients undergoing minimally invasive esophagectomy, the purpose of this study is to assess whether there is a potential advantage to receiving jejunostomy feedings for postoperative patients undergoing McKeown MIE as compared to the conventional nasoenteric tube feeding method.

DETAILED DESCRIPTION:
Esophageal cancer ranks ninth globally in terms of cancer incidence and sixth in terms of cancer deaths. In addition to the tumor itself and the surgical strike, nutrition and complications are two key factors limiting the rapid recovery of esophagectomy patients. A large number of studies have shown that rational nutritional support will help to improve the nutritional status of postoperative patients and reduce the risk of complications, and compared with parenteral nutrition, enteral nutrition has the advantages of lower complication rate, more economical and safer. Therefore, enteral nutrition is often recommended for esophageal cancer patients in the early postoperative period.

However, the commonly used clinical enteral nutrition includes transoral, nasoenteric tube (NT), gastrostomy and jejunostomy tube (JT) feeding. The optimal method of enteral nutrition after esophageal cancer surgery has been hotly debated in various published articles, but contradictions still exist. There have been numerous studies in recent years on the routine placement of jejunostomy tubes after esophageal cancer surgery, but none of them has yet reached an unanimously accepted conclusion.

Theoretically, a JT reduces the risk of detachment compared with an NT because the catheter is sutured to the abdominal wall; at the same time, a JT is placed deeper than an NT and farther away from the pyloric inlet, thus reducing the incidence of reflux. Most importantly, jejunostomy is considered to be comfortable and effective for long-term nutritional support, and patients can achieve long-term tube feeding at home through the JT, which can satisfy early discharge in case of insufficient oral intake and prevent readmission due to insufficient transoral intake.

Some studies have also confirmed these views, claiming that jejunostomy does not increase the incidence of total complications but improves QOL scores and short-term nutritional indices. It also eliminates the foreign body sensation of nasal mucosal nutritional tubes, and these patients showed acceptable tolerance to catheter insertion. Some researchers have also shown that jejunostomy does not affect the long-term oncological outcomes of patients undergoing esophageal cancer surgery, while increasing the incidence of perioperative complications, with data showing an overall complication rate of 13-38% after jejunostomy, and 0-3% of patients experiencing serious complications that require management, and therefore is not routinely recommended.

In summary, the final conclusion of the current clinical studies on whether to adopt jejunostomy after esophageal cancer resection is still controversial. Meanwhile, to the best of our knowledge, no study has yet examined the circumstances under which the option of performing a jejunostomy may be beneficial to patients. Therefore, in this study, on the basis of analyzing the relationship between the routine placement of jejunostomy tubes and tumor outcomes, and investigating whether jejunostomy brings benefits to patients after esophageal cancer surgery, we propose to conduct subgroup analyses of OS to clarify whether it may bring clear benefits to patients under certain circumstances, so as to guide clinicians to choose to perform this procedure in an appropriate manner.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients with a clear pathologic diagnosis of esophageal squamous cell carcinoma; 2. Received minimally invasive McKeown procedure; 3. Patients with R0 resection (R0: radical resection).

Exclusion Criteria:

* 1. Biopsy pathologic diagnosis of other types of esophageal cancer, e.g., adenocarcinoma; 2. Simultaneous combination of other primary cancers or history of other cancers; 3. Received minimally invasive Ivor-Lewis procedure or Sweet procedure; 4. Patients with R1 or R2 resection (R1 resection: microscopic tumor residue; R2: naked eye tumor residue); 5. Preoperative distant metastases; 6. Preoperative serious comorbidities in other systems; 7. Incomplete medical record data.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with EC who attended the Department of Thoracic Surgery at Daping Hospital and underwent the McKeown MIE procedure performed by the same surgical team were included for evaluation from September, 2017, to September, 2021.
Sampling Method: Non-Probability Sample
Enrollment: 577 (Actual)
Dates: Start 2023-12-13 (Actual); Primary Completion 2023-12-25 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
postoperative adverse events | Within 90 days after surgery
  including pneumonia, adult respiratory distress syndrome (ARDS), anastomotic leak (AL), vocal cord paralysis, chylothorax, pneumothorax, pleural effusion, cardiovascular complications
perioperative 90-day mortality. | Within 90 days

SECONDARY OUTCOMES:
Albumin loss rate | 7-10 days after surgery
  ((Preoperative albumin-POD7~10 albumin))⁄(Preoperative albumin) *100%

CONTACTS AND LOCATIONS:
Locations (1):
- Army Medical Center of the People's Liberation Army, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pu XS, Bao T, Wang YJ, Li KK, Yang Q, He XD, He Y, Yu J, Xie XF, Chen X, Guo W. Laparoscopic jejunostomy during McKeown minimally invasive esophagectomy: a propensity score analysis. Surg Endosc. 2025 Mar;39(3):1801-1810. doi: 10.1007/s00464-024-11519-x. Epub 2025 Jan 17. PMID 39821455